CLINICAL TRIAL: NCT04106323
Title: A Study of Factor Inhibitors in Adult Patients With Hemophilia and Von Willebrand's Disease in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Safaa AA Khaled (Other)
Responsible Party: Sponsor-Investigator, Safaa AA Khaled, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: SKhaled20
Record Dates: First submitted 2019-09-19; First posted 2019-09-27 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2019-10

CONDITIONS: Hemophilia; Von Willebrand Diseases; Christmas Disease
Keywords: Upper Egypt; Factor; Inhibitor
MeSH Terms: conditions — Hemophilia A; von Willebrand Diseases; Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemophilia A and B are bleeding disorders caused by deficiency of factor VIII and IX, respectively. The deficiency of one of these coagulation factors is due to a mutation on the X chromosome. Accordingly replacement of the deficient factor is currently the main treatment for these disorders. The most disappointing complication of replacement therapy in hemophilia is the development of inhibitors. Unlike haemophilia , inhibitor development in patients with V Willebrand's Disease (VWD) is a rare complication of treatment. Studies on inhibitors whether on hemophilia or VWD are limited in our region.

This study aims to

1. To estimate the frequency of factor inhibitors in hemophilia and VWD patients in our region.
2. To investigate modifiable risk factors associated with development of inhibitors in both diseases.
3. To correlate the level of inhibitor with the clinical presentation of the patients.
4. To assess influence of factor inhibitors on quality of life in patients who developed factor inhibitors in both diseases.

DETAILED DESCRIPTION:
Individuals with hemophilia are deficient in one of the clotting factor proteins that are vital in the formation of a clot. Classic hemophilia or hemophilia A is a deficiency of factor VIII, while Christmas Disease or Hemophilia B is a deficiency of factor IX. The prevalence of hemophilia A or B varies in different countries and geographic regions.

Patients with either type of hemophilia are at risk for prolonged bleeding, replacement of the deficient protein is the main therapy . The most serious complication of replacement therapy in hemophilia is the development of inhibitors.An inhibitor is a polyclonal high-affinity immunoglobulin G (IgG) that is directed against the clotting factorI protein. These antibodies can be either inhibitory or non inhibitory.

Inhibitors neutralize the administered clotting factor so that bleeding does not stop. Inhibitors are the most significant risk factor for morbidity and mortality associated with hemophilia, and patients with inhibitors present complex patient management challenges.

Few studies investigated development of factor inhibitor in Egyptian patients, however most of them concentrated on pediatric patients, also data regarding factor inhibitors in Upper Egypt was limited.

VonWillebrand's disease is a bleeding disorder caused by deficiency of VWF. The treatment of VWD is somewhat similar to that of patients with hemophilia which consists of infusions to replace the missing factors as on demand regimen using plasma derived (PD) products which contains both FVIII and VWF. Furthermore, many of the patients are currently on some form of prophylaxis to eliminate or decrease the frequency of bleeding episodes.

Nearly, 7.5 % of VWD patients develop inhibitors to VWF becoming non- responsive to replacement therapy, and prone to develop severe anaphylactic and life threatening reactions when exposed to any product that contains VWF.

Unlike hemophilia clinical presentation of VWD patients who developed inhibitors is not serious.

Again data on factor inhibitors in VWD is deficient in many countries worldwide particularly Egypt . Investigators assumed that this is the first study that well assess factor inhibitors in VWD in Upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed congenital hemophilia A, Christmas disease, and VWD

Exclusion Criteria

* Patients diagnosed with acquired hemophilia
* Patients below 18 years
* Patients with other bleeding tendencies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with hemophilia A, B, and Von willebrand's disease who will be admitted at the clinical hematology unit ( Department of Internal Medicine), Assiut University Hospital over one year will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2020-11-10 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with inhibitors | 4-days
  Frequency of inhibitors among patients with hemophilia A and B, and VWD
Number of patients on demand replacement therapy | 7-days
  Identification of the relationship between on demand replacement therapy and development of factor inhibitors in the study patients
Number of participants with low or high responding inhibitors | 7-days
  This would be assessed by of the relationship between inhibitor level and severity of clinical presentation of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Howaida A. Nafady, Prof., Study Director — Assiut University Hospial

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witmer C, Young G. Factor VIII inhibitors in hemophilia A: rationale and latest evidence. Ther Adv Hematol. 2013 Feb;4(1):59-72. doi: 10.1177/2040620712464509. PMID 23610614
- [Background] Ghosh K, Shukla R. Future of Haemophilia Research in India. Indian J Hematol Blood Transfus. 2017 Dec;33(4):451-452. doi: 10.1007/s12288-017-0862-4. Epub 2017 Aug 21. No abstract available. PMID 29075053
- [Background] Schep SJ, Boes M, Schutgens REG, van Vulpen LFD. An update on the 'danger theory' in inhibitor development in hemophilia A. Expert Rev Hematol. 2019 May;12(5):335-344. doi: 10.1080/17474086.2019.1604213. Epub 2019 Apr 25. PMID 30951401
- [Background] Hay CR, Palmer B, Chalmers E, Liesner R, Maclean R, Rangarajan S, Williams M, Collins PW; United Kingdom Haemophilia Centre Doctors' Organisation (UKHCDO). Incidence of factor VIII inhibitors throughout life in severe hemophilia A in the United Kingdom. Blood. 2011 Jun 9;117(23):6367-70. doi: 10.1182/blood-2010-09-308668. Epub 2011 Apr 6. PMID 21471523
- [Background] Hay CR, DiMichele DM; International Immune Tolerance Study. The principal results of the International Immune Tolerance Study: a randomized dose comparison. Blood. 2012 Feb 9;119(6):1335-44. doi: 10.1182/blood-2011-08-369132. Epub 2011 Nov 18. PMID 22101900
- [Background] Gouw SC, van den Berg HM, Oldenburg J, Astermark J, de Groot PG, Margaglione M, Thompson AR, van Heerde W, Boekhorst J, Miller CH, le Cessie S, van der Bom JG. F8 gene mutation type and inhibitor development in patients with severe hemophilia A: systematic review and meta-analysis. Blood. 2012 Mar 22;119(12):2922-34. doi: 10.1182/blood-2011-09-379453. Epub 2012 Jan 26. PMID 22282501
- [Background] Peyvandi F, Mannucci PM, Garagiola I, El-Beshlawy A, Elalfy M, Ramanan V, Eshghi P, Hanagavadi S, Varadarajan R, Karimi M, Manglani MV, Ross C, Young G, Seth T, Apte S, Nayak DM, Santagostino E, Mancuso ME, Sandoval Gonzalez AC, Mahlangu JN, Bonanad Boix S, Cerqueira M, Ewing NP, Male C, Owaidah T, Soto Arellano V, Kobrinsky NL, Majumdar S, Perez Garrido R, Sachdeva A, Simpson M, Thomas M, Zanon E, Antmen B, Kavakli K, Manco-Johnson MJ, Martinez M, Marzouka E, Mazzucconi MG, Neme D, Palomo Bravo A, Paredes Aguilera R, Prezotti A, Schmitt K, Wicklund BM, Zulfikar B, Rosendaal FR. A Randomized Trial of Factor VIII and Neutralizing Antibodies in Hemophilia A. N Engl J Med. 2016 May 26;374(21):2054-64. doi: 10.1056/NEJMoa1516437. PMID 27223147
- [Background] Miller CH, Platt SJ, Rice AS, Kelly F, Soucie JM; Hemophilia Inhibitor Research Study Investigators. Validation of Nijmegen-Bethesda assay modifications to allow inhibitor measurement during replacement therapy and facilitate inhibitor surveillance. J Thromb Haemost. 2012 Jun;10(6):1055-61. doi: 10.1111/j.1538-7836.2012.04705.x. PMID 22435927
- [Background] Soucie JM, Miller CH, Kelly FM, Payne AB, Creary M, Bockenstedt PL, Kempton CL, Manco-Johnson MJ, Neff AT; Haemophilia Inhibitor Research Study Investigators. A study of prospective surveillance for inhibitors among persons with haemophilia in the United States. Haemophilia. 2014 Mar;20(2):230-7. doi: 10.1111/hae.12302. Epub 2013 Nov 22. PMID 24261612
- [Background] Duncan E, Collecutt M, Street A. Nijmegen-Bethesda assay to measure factor VIII inhibitors. Methods Mol Biol. 2013;992:321-33. doi: 10.1007/978-1-62703-339-8_24. PMID 23546724
- [Background] Pokras SM, Petrilla AA, Weatherall J, Lee WC. The economics of inpatient on-demand treatment for haemophilia with high-responding inhibitors: a US retrospective data analysis. Haemophilia. 2012 Mar;18(2):284-90. doi: 10.1111/j.1365-2516.2011.02623.x. Epub 2011 Aug 4. PMID 21812862